CLINICAL TRIAL: NCT05517369
Title: Impact of Using Hybrid-ESD+ and LiftUp® as Injectable on en Bloc/R0 Rate in Colorectal Adenomas Between 2 and 3 cm.
Brief Title: Impact of Hybrid-ESD+ and LiftUp® on the en Bloc/R0 Rate in Colorectal Adenomas Between 2 and 3 cm
Acronym: HADRIAN
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants fitting into the study
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: Waid City Hospital, Zurich (Other); University Hospital Ulm (Other); Rems-Murr-Klinikum Winnenden (Unknown); Insel Gruppe AG, University Hospital Bern (Other); Klinikum Ludwigsburg (Other); Mathilden Hospital Herford (Unknown); St. Franziskus Hospital Münster (Unknown); Agaplesion Kliniken Kassel (Unknown); Ovesco Endoscopy AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Brand_HADRIAN_10_08_2022; WHO Universal Trail Number (Other: U1111-1281-5357)
Record Dates: First submitted 2022-08-12; First posted 2022-08-26 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Colorectal Adenoma
Keywords: Hybrid-ESD+; Endoscopic Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hybrid-ESD+ (Experimental): All participants receive resection of non-pedunculated colorectal polyp between 2 and 3 cm using the Hybrid-ESD+ method.
  Interventions: Procedure: Hybrid ESD+

INTERVENTIONS:
Procedure: Hybrid ESD+ — Injection of the Lift Up solution, followed by circumcision of the lesion using a snare tip or ESD knife. Using an additional working channel (AWC), the lesion is resected using a grasper and snare.

SUMMARY:
This study examines whether the use of Hybrid-ESD+ with LiftUp (Injection solution) results in a higher en bloc and/or R0 rate for non pedunculated colorectal adenomas between 2 and 3 cm than described in the literature for conventional EMR.

DETAILED DESCRIPTION:
There are several options for endoscopic polypectomy of polyps between 2-3 cm, all of which have their advantages and disadvantages and none of which has yet become the established standard procedure.

Conventional EMR has the disadvantage of more frequent residuals and/or recurrences due to lack of en bloc resection, while ESD has the disadvantage of being more complex and complications more likely.

A possible alternative is the use of hybrid ESD+ with LiftUp subcutaneous injection. The method with the LiftUp gel forming a stable gel cushion under the lesion, in combination with the circular circumcision of the mucosa at this site and the AWC for the current loop and the grasper, could achieve a better en bloc resection rate with a low complication rate than other procedures mentioned above.

The higher effectiveness in terms of recurrences and complications could subsequently result in a reduction of endoscopic or surgical re-interventions.

In this study, non-pedunculated colorectal polyps between 2 and 3cm in size are resected using ESD+ method and lift up as an injection solution.

Methodological and clinical parameters are recorded. After 4 weeks, the patients are contacted by telephone to record possible late effects.

If an endoscopic control is performed after 6 months (according to the guideline or according to the investigator), the findings are also recorded.

ELIGIBILITY:
Inclusion Criteria:

* Non-pedunculated lesion in the colorectum (epithelial lesion, 2-3 cm).
* Ablation medically indicated and possible (coagulation, etc. - as determined by the center)

Exclusion Criteria:

* Age < 18 years
* Pedunculated lesion (Paris0-Ip)
* Size of the lesion <2cm or >3cm
* Pregnant and breastfeeding women
* Patient not capable of informed consent / consent not possible
* Bioptic evidence of a carcinoma / high probability of the presence of a carcinoma
* Non-lifting sign / known recurrence after previous therapy
* Impassable stenosis in the colon / rectum
* Patients with compelling need for therapeutic anticoagulation or dual antiplatelet therapy that cannot be discontinued for resection
* As per contraindications from the AWC & LiftUp Instructions for Use:
* The AWC is not to be used if flexible-endoscopic procedures are contraindicated.
* The LiftUp gel should not be used when flexible endoscopic procedures are contraindicated, especially in combination with submucosal endoscopic resection (EMR) or endoscopic submucosal dissection (ESD) injectables.
* LiftUp gel should not be used in patients with known sensitivity to any of the ingredients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate of non pedunculated colorectal polyps between 2 and 3cm using hybrid ESD+ | after 14 days
  In how many cases a complete R0 resection (basal and lateral margin) is found on pathologic examination

SECONDARY OUTCOMES:
Complication rate (perforations, bleeding) | up to 4 weeks
  Perforation: dehiscence of the muscularis propria diagnosed during or after resection.
  Hemorrhage:
  * Clinically significant post-endoscopic bleeding (CSPEB). Bleeding from the ablation site with hematochezia after completion of index colonoscopy
  * Intraprocedural bleeding (IPB). Percent, defined as bleeding lasting > 60 seconds during intervention necessitating therapy
Recurrence rate | 6 months
  Rate of adenoma residue and/or adenoma recurrence in percent after 6 months. This is determined by the colonoscopic and histologic findings from 2 biopsies from the scar or resection specimen.
Procedural parameters - Intervention duration | 1 day
  Intervention duration (time range from injection to complete resection)
Procedural parameters - Cleanliness of the colon | 1 day
  Cleanliness of the colon (according to the Boston Bowel Preparation Scale (BBPS) 0-9)
Localization of polyp | 1 day
  Position of the polyp within the colon (Coecum, Ascendens, Transversum, Deschendens, Sigmoid, Rectum)
Polyp size | 1 day
  Polyp diameter in mm
Polyp morphology | 1 day
  according to paris classification
Polyp histology | 7 days
  histological examination (tubular, tubulovillous, villous)
Duration of hospital stay | up to 4 weeks
  Time frame from first day to discharge

CONTACTS AND LOCATIONS:
Locations (9):
- Germany (7):
  - Mathilden Hospital Herford, Herford
  - Agaplesion Diakonie Kliniken Kassel, Kassel
  - Klinikum Ludwigsburg, Ludwigsburg
  - St. Franziskus Hospital Münster, Münster
  - Universitätsklinikum Ulm, Ulm
  - Rems-Murr-Klinikum Winnenden, Winnenden
  - Universitätsklinik Würzburg, Würzburg
- Switzerland (2):
  - Inselspital Bern, Bern
  - Stadtspital Waid, Zurich

IPD SHARING:
Plan to Share IPD: No